CLINICAL TRIAL: NCT00594828
Title: Randomized Controlled Trial of Patient Self-Testing of Warfarin Therapy Using an Internet Based Expert System
Brief Title: Patient Self Testing of Warfarin Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College Cork (Other)
Collaborators: Hoffmann-La Roche (Industry); Health Research Board, Ireland (Other); ZyCare Inc (Industry)
Responsible Party: Dr Susan O'Shea, University College Cork
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PA/05/16
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Warfarin
Keywords: Patient self-testing; Oral anticoagulation therapy; Expert Systems; Point-of-Care Systems; International Normalized Ratio

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): 6 months of supervised patient self testing using an expert system
  Interventions: Device: CoaguChek (Patient self testing)
- 2 (Active Comparator): 6 months of routine medical care by the anticoagulation management service
  Interventions: Device: Anticoagulation Management Service (AMS)

INTERVENTIONS:
Device: CoaguChek (Patient self testing) — Patients will test their INR at home either biweekly, weekly or every 2 weeks using a CoaguChek point of care meter and communicate with the healthcare provider via an internet based expert system
  Other Names: CoaguChek S point of care meter; CoaguChek XS point of care meter; CoagCare expert system
  Arms: 1
Device: Anticoagulation Management Service (AMS) — Patients will attend the AMS for six months and have their INR checked every 4-6 weeks or more frequently, at the discretion of the clinician
  Arms: 2

SUMMARY:
To test the hypothesis that home international normalised ratio (INR) monitoring with supervised patient self-testing (PST)can provide comparable or superior time in therapeutic range (TTR) to that provided by traditional outpatient anticoagulation.

DETAILED DESCRIPTION:
Indications for anticoagulant treatment to prevent thromboembolic disease have increased in recent years. INR must be monitored frequently to determine the safest dose and to minimize the risk for thrombotic and haemorrhagic complications. Standard warfarin therapy is associated with rates of major haemorrhage of up to 5-9% annually and recurrent venous thromboembolism of up to 8%. These event rates are dependent of the model of care used to manage warfarin therapy, with better outcomes associated with home testing of the INR which enables patients to monitor their response to warfarin more frequently. INR results must still be 'managed' by communicating the data to the healthcare provider, usually be telephone or fax.

In this study we will evaluate a novel method of PST; supervised PST with an internet based expert system, which 'manages' patients on oral anticoagulation by utilizing clinical and laboratory data provided by the patient and dose adjustment and retesting algorithms derived from clinical practice. Patients will be randomized to either 6 months of supervised PST or routine medical care by the AMS. At the end of the 6 month period, each patient will then 'cross over' to the other management regimen and the difference in TTR between the two periods will be compared.

ELIGIBILITY:
Inclusion Criteria:

* on warfarin therapy for a minimum of 2 months
* are expected to be on warfarin therapy for the duration of the 12 month study
* internet access

Exclusion Criteria:

* inability to provide informed consent
* inability to use a home INR meter
* patients who do not have a telephone
* more than 2 missed clinic appointments in the preceding 6 months
* patients on anticoagulant drugs other than warfarin (eg heparin, low molecular weight heparin)
* history of hemorrhagic complications with a therapeutic or therapeutic INR in the preceding 6 months
* inability to attend the hospital at short notice, if necessary

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2006-07; Primary Completion 2009-04 (Estimated); Study Completion 2008-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome variable used to assess therapeutic efficacy and safety will be the difference in TTR during the six months of AMS management and the six months of PST | 1 year

SECONDARY OUTCOMES:
To compare the number of adverse events (haemorrhagic and thromboembolic) using PST and AMS management | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Susan J O'Shea, MD, Principal Investigator — Cork University Hospital
Locations (1):
- Cork University Hospital, Cork, Cork, Ireland